CLINICAL TRIAL: NCT04775498
Title: Non-inferiority Study Comparing Two Psychoeducation Programmes (Mobile Application Versus Face-to-face Psychoeducation Group) in a Population of Patients With Bipolar Disorder
Brief Title: Psychoeducation Programmes - Patients With Bipolar Disorder
Acronym: AppEduc-BD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PREPS 2017 SAMALIN
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder Type I or II (According to DSM-5)
Keywords: Bipolar disorder; Psychoeducation; Mobile application; Smartphone; Recurrence prevention
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: * Standard group : patients will participate at all sessions of face-to-face psychoeducation (sessions labeled and controlled by their Regional Health Agency).
  * Experimental group: patients will use SIMPLe application during 12 months.
Masking Description: Eligible patients after obtaining their consent will be randomized:
  * either in the face-to-face psychoeducation group and will benefit from a programme of psychoeducation sessions available at the participating center.
  * or in the SIMPLe application group and will have access to the application (personal access).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face psychoeducation group (Active Comparator): The group of face-to-face psychoeducation or standard intervention will consist of the participation by the patients include in all the sessions of a therapeutic education programme of the investigator center.
  Interventions: Behavioral: Face-to-face psychoeducation group
- SIMPLe mobile application (Experimental): The experimental intervention consists of the use of the SIMPLe application during 1 year: answers of 5 daily questions and to the weekly questions. Moreover, daily and personalized psychoeducation messages (adapted to the answers to the tests carried out) will be sent to user by notifications.
  Interventions: Behavioral: SIMPLe mobile application

INTERVENTIONS:
Behavioral: Face-to-face psychoeducation group — All of the investigation centers participating in this study have a psychoeducation programme on bipolar disorders labeled and monitored by their Regional Health Agency. For this, he must respect the decree of January 14, 2015 relating to the specifications of therapeutic education programs for the patient. Patients will be receive by an investigator, for inclusion and baseline evaluation and at 6 and 12 months after inclusion. During this meeting, investigator and patient will be complete 7 questionnaires (about disease, treatment observance and quality of life), investigator will collect treatment, style life and adverse event(s).
  Arms: Face-to-face psychoeducation group
Behavioral: SIMPLe mobile application — The experimental intervention consists of 12 months use SIMPLe smartphone application who has been developed by the Barcelona Institute of neuroscience. The purpose of this application is to deliver individualized psychoeducation messages to the patient's clinical condition. The psychoeducational messages correspond to the contents of the different modules and sessions carried out in face-to-face psychoeducation groups (Colomm & Vieta ; 2015). Patients will be receive by an investigator for inclusion and baseline evaluation, at 6 and 12 months after inclusion. During this meeting, investigator and patient will be complete 7 questionnaires (about disease, treatment observance and quality of life), investigator will collect treatment, style life and adverse event(s).
  Arms: SIMPLe mobile application

SUMMARY:
This is a controlled, randomized, prospective, open-label, non-inferiority trial lasting 12 months. The effectiveness of using a psychoeducational smartphone application (SIMPLe) will be compared to the effectiveness of face-to-face group psychoeducation.

DETAILED DESCRIPTION:
Bipolar disorder (affecting 3 to 5% of French population) is characterized by the recurrence of severe symptomatic periods (depression, mania, hypomania) and interepisodic periods characterized by the persistence of residual symptoms, impaired psychosocial functioning and quality of life. The combination of psychosocial strategies with drug treatment is associated with an improvement in the prognosis of the disease. Among these complementary strategies, psychoeducation has been shown to be effective in reducing the risk of recurrence, the length of hospital stays and improving compliance. It improves an individual's understanding and knowledge of their disorder and its various treatments. Despite its effectiveness, psychoeducation for bipolar disorder remains relatively scarcely applied in France due to a limited healthcare offer (44 available programmes labeled by the Regional Health Agencies in 2017).

In recent years, a significant number of smartphone applications have been developed in the field of mental health. To date, none of these applications has proven effective in patients with bipolar disorder. In this context, the Institute of Neuroscience of Barcelona has developed a "SIMPLe" application to assess and record a subject's symptoms and deliver personalized psychoeducation. In terms of efficacy, a study has shown the interest of this application in improving biological rhythms, thereby reducing the risk of relapse and improving psychosocial functioning and the quality of life of patients suffering from bipolar disorder in remission phase. This application has been translated and adapted into French as part of a partnership with the Barcelona Institute of Neuroscience. However, the benefits of this type of application in terms of effectiveness, accessibility or reduction of health costs have never been studied in comparison to face-to-face psychoeducation programmes. This research project therefore represents a real opportunity to evaluate for the first time the effectiveness of an application allowing the delivery of personalized psychoeducation in comparison to a face-to-face group psychoeducation program (reference treatment for relapse prevention).

The SIMPLe app includes 5 daily questions (mood, energy, sleep, irritability, medication adherence) that will assess different areas associated with bipolar disorder. The user will also receive a weekly test to determine the presence and intensity of depressive or manic symptoms. Daily and personalized psychoeducation messages (adapted to the answers to the tests carried out) will be sent to the user by notifications. The app contains a bank of around 400 psychoeducational messages, based on Prof. Vieta and Dr Colom's Psychoeducation Manual for Bipolar Disorders.

Eligible patients, after obtaining their consent, will be randomized (i) either in the face-to-face psychoeducation group which will consist of the participation by the patients in all the sessions of a therapeutic education program (labeled and controlled by their Regional Health Agency) of the investigator center, (ii) or in the SIMPLe application group and will benefit from access to the application via a code that will be sent to them.

Three additional visits to the usual care are planned (assessment visit, 6 months and 12 months). At each visit, patients must complete questionnaires (CSRI, YMRS, MADRS, FAST, MARS, WHOQOL-BREF and EQ-5D).

The hypothesis formulated by the investigator is that a psychoeducational strategy using the SIMPLe smartphone application has an effect comparable to participation in a face-to-face psychoeducation group, in term of the recurrence prevention in a sample of stabilized patients with bipolar disorder (at 12 months). The recurrence rate is defined by the percentage of patients having presented a mood episode of bipolar disorder, namely a major depressive episode, manic or hypomanic episode, according to the criteria of DSM-5 and on the basis of the judgment of the clinician since the beginning of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from bipolar disorder (type 1 or 2) according to DSM-5 criteria
* Not presenting a mood episode according to DSM-5 criteria
* Stable for at least 1 month with scores on YMRS < 8 and MADRS < 8
* Owning a smartphone
* Agreeing to attend group psychoeducation sessions
* Having no problem understanding fluent French
* Having given free and informed consent and signed the consent to participate in the study
* Available for 12 onth follow-up

Exclusion Criteria:

* Not having a smartphone compatible with the SIMPLe application
* Cannot attend psychoeducation group sessions on a regular basis
* Not having given their consent to participate in the study or unable to give their informed consent
* Not affiliation with a social security scheme
* Having a legal protection measure (safeguard of justice or guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 12 months after inclusion
  Measure the difference of recurrence rate (defined by the percentage of patients having presented a mood episode of bipolar disorder, namely a major depressive episode, manic or hypomanic episode, according to the criteria of DSM-5 and on the judgment of the clinician since the beginning of the intervention) between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application

SECONDARY OUTCOMES:
Hospitalization number | 6 months after inclusion
  Measure the difference of number and duration of hospitalization between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application
Hospitalization number | 12 months after inclusion
  Measure the difference of number and duration of hospitalization between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application
Maniac and depressive symptomatology intensity | 6 months after inclusion.
  Measure the difference of maniac and depressive symptomatology intensity between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. These measures are based on YMRS (for maniac symptomatology) questionnaire.
Maniac and depressive symptomatology intensity | 12 months after inclusion.
  Measure the difference of maniac and depressive symptomatology intensity between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. These measures are based on YMRS (for maniac symptomatology) questionnaire.
Maniac and depressive symptomatology intensity | 6 months after inclusion.
  Measure the difference of maniac and depressive symptomatology intensity between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. These measures are based on MADRS (for depressive symptomatology) questionnaires.
Maniac and depressive symptomatology intensity | 6 months after inclusion.
  Measure the difference of medication compliance between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on MARS (Medication Adherence Report Scale) questionnaire.
Medication compliance | 12 months after inclusion.
  Measure the difference of medication compliance between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on MARS (Medication Adherence Report Scale) questionnaire.
Psychosocial functioning | 6 months after inclusion.
  Measure the difference of psychosocial functioning between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on FAST (Functional Analysis Screening Tool ) questionnaire.
Psychosocial functioning | 12 months after inclusion.
  Measure the difference of psychosocial functioning between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on FAST (Functional Analysis Screening Tool ) questionnaire.
Evaluation of Quality of life | 6 months ater inclusion
  Measure the difference of quality of life between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on WHOQOL-BREF (World Health Organization Quality of Life) questionnaire.
Evaluation of Quality of life | 12 months ater inclusion
  Measure the difference of quality of life between patients who participated to face-to-face psychoeducation group and patients who use SIMPLe application. This measure is based on WHOQOL-BREF (World Health Organization Quality of Life) questionnaire.
Cost efficiency | 12 month after inclusion
  Cost efficiency evaluation of SIMPLe application using CSRI (Client Service Receipt Inventory) questionnaire
Cost / utility ratio | 12 month after inclusion
  Evaluation of cost / utility ratio of SIMPLe application using the EQ-5D (EuroQol 5 Dimensions) questionnaire.
Qualitative analysis | 12 months after inclusion
  Some patients of SIMPLe application group (4 womens and 4 mens < 30 years, 4 womens and 4 mens 30 to 50 years and 4 womens and 4 mens > 50 years) will participate in an individual interview. These semi-structured individual interviews will be carried out by a psychologist. During these interviews the perception and use of the SIMPLe application by patients will be gathered (both positive opinions and negative criticisms and possible obstacles to its use).

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic Samalin, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (10):
- France (10):
  - CH Charles Perrens, Bordeau
  - CHU - Gabriel Montpied, Clermont-Ferrand
  - CHU - Hôpital Lapeyronie, Montpellier
  - CHU, Nantes
  - CHU - Hôpital Universitaire Carémeau, Nîmes
  - APHP - Hôpital Fernand-Widal, Paris
  - CH Saint-Anne, Paris
  - APHP - Centre Hospitalier Henri Mondor, Paris
  - CHI HC site rives du Doubs Pontarlier, Pontarlier
  - CHU - Hôpital de Psychiatrie, Toulouse